CLINICAL TRIAL: NCT06064929
Title: An Open Label Phase 1b Study of Felzartamab in Lupus Nephritis
Brief Title: A Study to Learn More About the Safety and Effects of Felzartamab in Adults With Lupus Nephritis Aged 18 to 75 Years Old
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HI-Bio, A Biogen Company (Industry)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 299LE101; HIB-202-101 (Other: Human Immunology Biosciences (HI-Bio))
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis
Keywords: Felzartamab; LN; Systemic Lupus Erythematosus; Lupus; Refractory LN
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — felzartamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Felzartamab (Experimental): Participants will receive two courses of multiple intravenous (IV) doses of felzartamab, separated by a 28-week off-treatment period.
  These courses are given in Part 1 and Part 2 of the trial.
  Interventions: Drug: Felzartamab

INTERVENTIONS:
Drug: Felzartamab — Administered IV
  Other Names: HIB202; BIIB148; MOR202; MOR03087; TJ202

SUMMARY:
In this study, researchers will learn more about the use of felzartamab in people with active lupus nephritis, also known as LN. In people with LN, antibodies build up in the glomeruli of the kidneys. Antibodies are proteins in the blood used by the immune system to fight infection. Glomeruli are small filters that remove waste and extra fluid from the blood. This buildup leads to inflammation and damage to the kidneys.

Kidney damage can lead to too much protein and blood leaking into the urine. High levels of protein in the urine, called proteinuria, are common in people with LN. Symptoms of LN can include fever, swelling in the legs and body, and high blood pressure. If left untreated, LN can eventually lead to kidney failure.

In this study, researchers will learn more about how a study drug called felzartamab affects people with LN. Felzartamab is a monoclonal antibody, which means it is an antibody made in a laboratory. Felzartamab can target immune cells that produce antibodies, helping to lower their buildup in the kidneys. The main goal of this study is to learn more about the safety of felzartamab and how it works in the body of people with LN who are taking standard of care. This will help researchers decide if they should do more studies with felzartamab in people with LN. Standard of care is the usual treatment or care given to patients for a disease, as prescribed by their doctor.

The main question researchers want to answer in this study are:

• How many participants had adverse events during the study? An adverse event is a health problem that may or may not be caused by the study drug. It can happen during a clinical study or within a certain amount of time after the study has ended.

Researchers will also learn more about:

* How much felzartamab affects proteinuria and the level of creatinine in the urine. Creatinine is a protein that is released into the blood from normal muscle wear and tear. Its levels can help doctors understand how well your kidneys are working.
* How many participants have a complete response. A complete response means that their urine protein levels decrease to a low level, and their kidney function stays stable.
* How many participants have a 50% decrease in the level of protein and creatinine in their urine.
* How much felzartamab affects the participants' lupus-related blood tests.
* How the body processes felzartamab.
* How many participants develop antibodies against felzartamab in the blood.

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 42 days.
* Throughout the study, all participants will continue taking their standard of care, as prescribed by their doctor.
* There are 2 parts in this study. In both parts, participants will receive felzartamab through an intravenous infusion, also known as an IV. This means it is being given into a vein.
* In Part 1, participants will have up to 14 visits to their study research center. In Part 2, participants may have up to 15 visits.
* Each participant will be in the study for about 2 years.

DETAILED DESCRIPTION:
Study Sponsor, originally HI-Bio, Inc., is now HI-Bio, A Biogen Company.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Diagnosis of Systemic Lupus Erythematosus (SLE) according to the 2019 European League Against Rheumatism (EULAR)/ American College of Rheumatology (ACR) criteria
* Diagnosis of International Society of Nephrology/ Renal Pathology Society (ISN/RPS) 2003 Class III or IV LN as evidenced by renal biopsy performed within 1 year prior to or during screening, either with or without the presence of Class V LN
* Proteinuria (urine protein to creatinine ratio) > 1.0 gram per gram (g/g), based on 24-hour urine collection during screening
* eGFR ≥ 45 milliliter/minute/1.73 square meters (mL/min/1.73 m^2) (as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula)

  1. If eGFR is ≥35 to <45 mL/min/1.73m^2, renal biopsy must be within 6 months of screening and must not have >50% of glomeruli with sclerosis. If the renal biopsy was performed more than 6 months prior to screening, a repeat biopsy must be done during screening after all the other eligibility criteria are met
  2. If eGFR is ≥45 mL/min/1.73 m^2, renal biopsy must be within 1 year prior to screening. If the renal biopsy was performed more than 1 year prior to screening, a repeat biopsy must be done during screening after all the other eligibility criteria are met
* History of inadequate response, for lack of efficacy or intolerance, to at least a three-month course of one standard of care treatment for lupus nephritis, as determined by the treating physician

Part 2

* Participants must complete Part 1 of the study to be eligible to participate in Part 2.

Exclusion Criteria:

Part 1

* Presence of rapidly progressive glomerulonephritis, as defined by at least one of the following: crescent formation in > 50% of glomeruli on renal biopsy, sustained doubling of serum creatinine within 12 weeks of screening, or the investigator's opinion that the participant has rapidly progressive glomerulonephritis
* Greater than 50% of glomeruli with sclerosis on renal biopsy
* Currently requiring hemodialysis or peritoneal dialysis or expected to require dialysis during the study treatment period
* A previous kidney transplant or other organ transplant, or planned transplant within study treatment period

Part 2

* Did not complete Part 1 of the study
* Received protocol-prohibited medications in Part 1 such as calcineurin inhibitors (e.g., cyclosporine, tacrolimus, or voclosporin), alkylating agents including cyclophosphamide, or biologic agents other than felzartamab
* Progression of LN (as measured by worsening proteinuria and/or decreasing eGFR) has been observed such that in the opinion of the investigator the participant will not benefit from continuing in Part 2 of the study

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to Week 104

SECONDARY OUTCOMES:
Change from Baseline in Urine Protein:Creatinine Ratio (UPCR) | Baseline, Up to Week 104
Proportion of Participants Who Achieve a Complete Renal Response (CRR) | Week 24
Proportion of Participants Who Achieve Overall Complete and Partial Renal Response (PRR: CRR+PRR) | Week 24
Change from Baseline in Serum Creatinine | Baseline, Up to Week 104
Change from Baseline in Urine Protein | Baseline, Up to Week 104
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Up to Week 104
Change from Baseline in eGFR Slope | Baseline, Up to Week 104
Change from Baseline in Lupus Serologic Markers | Baseline, Up to Week 104
Felzartamab Serum Concentrations | Up to Week 104
Number of Participants with Anti-drug Antibodies to Felzartamab | Baseline, Up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — HI-Bio, A Biogen Company
Locations (24):
- United States (14):
  - University of California, San Diego (UCSD), La Jolla, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - ClinCept, LLC/River City Vascular Specialists LLC, Columbus, Georgia
  - Georgia Nephrology - Lawrenceville, Lawrenceville, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Joseph S. and Diane H. Steinberg Ambulatory Care Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - Precision Comprehensive Clinical Research Solutions - Grapevine, Grapevine, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Accurate Clinical Research - Katy, Katy, Texas
  - R & H Clinical Research, Katy, Texas
- Argentina (3):
  - Hospital Britanico de Buenos Aires, Caba, Buenos Aires F.D.
  - CEMIC, CABA, Buenos Aires F.D.
  - Clinica Priv Velez Sarsfield, Córdoba, Córdoba Province
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Melbourne, Victoria
  - Western Health, Saint Albans, Victoria
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - University Health Network - Toronto General Division, Toronto, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/